CLINICAL TRIAL: NCT04473001
Title: Continuous Glucose Measurements to Detect Hypoglycemia in Patients Undergoing Major Surgery
Brief Title: Wireless Assessment of Respiratory and Circulatory Distress - Continuous Glucose Monitoring
Acronym: WARD-CGM
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Jakob Carlsson, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H-20002220
Record Dates: First submitted 2020-06-30; First posted 2020-07-16 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Hypoglycemia; Perioperative Complication
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical patients: Adult patients admitted for major abdominal-, orthopedic or arterial vascular surgery.
  Interventions: Other: Continuous vital signs and glucose monitoring

INTERVENTIONS:
Other: Continuous vital signs and glucose monitoring — The patients will have the following parameters and vital signs continuously monitored using wireless equipment:
  * Glucose measurements (quasi-continuous, every 5 minutes)
  * Heart rate
  * Heart rhythm (single-lead ECG; quasi-continuous, 10 seconds every minute)
  * Signs of cardiac ischemia (single-lead ECG; quasi-continuous, 10 seconds every minute)
  * Respiration rate
  * Oxygen saturation of arterial hemoglobin (%SpO2)
  * Perfusion index (ratio of the pulsatile blood flow to the non-pulsatile or static blood in peripheral tissue)
  * Blood pressure (quasi-continuous; every 30-60 minutes)
  * Skin temperature
  * Electrodermal activity
  * Ambulatory activity (accelerometry)

SUMMARY:
The applicant and research team partners have over the last years developed the WARD project (Wireless Assessment of Respiratory and circulatory Distress), using wireless continuous monitoring of vital signs in high-risk patients undergoing major abdominal surgery. An important perioperative indicator not currently included in the WARD project is continuous glucose monitoring (CGM), which may not only predict and identify hypo- and hyperglycemia, but also utilize the information from variations in blood glucose in combination with other changes in vital signs to predict surgical complications in all patients.

The current study involves the inclusion of 80 patients, scheduled for major abdominal, orthopedic or vascular surgery, to be monitored with CGM in addition to the currently measured vital signs. The project is a prospective, observational, clinical study, describing and analyzing variations in perioperative blood glucose levels and vital signs, and the relation to adverse clinical outcomes.

Patients scheduled for elective surgery will preferentially be recruited at the preoperative assessment at a maximum of 30 days before surgery. CGM and monitoring of the remaining vital sign modalities will commence on the day of surgery. Patients admitted for acute surgery will be recruited preoperatively and CGM as well monitoring of the remaining vital sign modalities will commence as soon as possible. The patients will be monitored with CGM for up to 10 days and with the remaining modalities for up to 5 days or for all modalities until discharge or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted to Rigshospitalet or Bispebjerg Hospital for major abdominal surgery (e.g. colonic resections, gastrectomy, hepatic resection etc.) or major orthopedic surgery (e.g. hip-fracture, hip and knee-arthroplasty) or major arterial vascular surgery (e.g. aortic aneurysm, iliac or femoral bypass etc.)
* Estimated duration of surgery ≥1 hour and at least one expected overnight stay postoperatively

AND

● Type 1 diabetes (Clinically defined: insulin initiated at diabetes onset and treatment with multiple doses of insulin or continuous subcutaneous insulin infusion) (n=20)

OR

● Type 2 diabetes treated with insulin (Clinically defined: treatment with diet or oral antidiabetic drugs for at least 6 months before insulin was started) (n =20)

OR

● Type 2 diabetes treated with oral antihyperglycemic drugs and/or GLP-1 analogs (n=20)

OR

● No diabetes mellitus (excluded by an admission HbA1c <48 mmol/mol) (n=20)

Exclusion Criteria:

* Patient expected not to cooperate with study procedures.
* Patient allergic to plaster or silicone.
* Patients with impaired cognitive function (assessed by a Mini Mental State Examination [MMSE] score <24)
* Patients admitted for palliative care only.
* Previous or currently scheduled for pancreatectomy (complete or partial)
* Patients with pacemaker or implantable cardioverter defibrillator (ICD) device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted for major abdominal-, orthopedic or arterial vascular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Duration of glucose levels < 3.9 mmol/L as measured by continuous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Active CGM | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  % of study time with active CGM and data stored on the secure server
Glycemic variability | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Glycemic variability (%CV, SD)
Mean glucose | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Mean glucose (mmol/L).
Number of hypoglycemic events | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Median number of hypoglycemic events per patient per day; glucose < 3.9 mmol/L, >15 minutes
Number of severe hypoglycemic events | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Median number of severe hypoglycemic events per patient per day; glucose < 3.0 mmol/L, >15 minutes
Number of fasting hypoglycemia events | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Median number of hypoglycemia events during perioperative fasting; glucose < 3.9 mmol/L, >15 minutes
Duration of fasting hypoglycemia events | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Duration of hypoglycemia events during perioperative fasting, glucose < 3.9 mmol/L
% of readings and time below range (TBR) | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  * % of readings and time in range 3.0-3.8 mmol/L
  * % of readings and time <3.0 mmol/L
% of readings and time in range (TIR) | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  ○ % of readings and time in range 3.9-10.0 mmol/L.
% of readings and time above range (TAR) | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  * % of readings and time in range 10.1-13.9 mmol/L.
  * % of readings and time >13.9 mmol/L.
Adverse clinical outcomes | Until 30 days after monitoring is commenced
  Occurrence and severity of a range of predefined adverse clinical outcomes.
Readmission or death | Until 6 months after monitoring is commenced
  Occurrence of readmission and/or death.

OTHER OUTCOMES:
Agreement between CGM and plasma glucose (PG) | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Level of agreement between CGM and concomitant PG measurements.
Duration of hypoglycemia as measured by PG | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Duration of glucose levels < 3.9 mmol/L as measured by plasma glucose (defined as time from first measurement < 3.9 mmol/L, until first measurement > 3.9 mmol/L).
Number of PG measurements | Through the monitoring period (up to 5 days after monitoring is commenced or until discharge)
  Median number of bedside PG measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, MD, DMSc, Study Director — Rigshospitalet, Centre for Cancer and Organ Diseases
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen, Danmark
  - Bispebjerg Hospital, Copenhagen, Danmark

REFERENCES:
- [Derived] Carlsson CJ, Norgaard K, Oxboll AB, Sogaard MIV, Achiam MP, Jorgensen LN, Eiberg JP, Palm H, Sorensen HBD, Meyhof CS, Aasvang EK. Continuous Glucose Monitoring Reveals Perioperative Hypoglycemia in Most Patients With Diabetes Undergoing Major Surgery: A Prospective Cohort Study. Ann Surg. 2023 Apr 1;277(4):603-611. doi: 10.1097/SLA.0000000000005246. Epub 2021 Oct 8. PMID 35129526